CLINICAL TRIAL: NCT02337205
Title: A Phase 1, Single-Center, Safety, Tolerability, and Pharmacokinetic Study of KX2 391 Ointment in Subjects With Actinic Keratosis
Brief Title: Ph 1, Single-Center, Safety, Tolerability & Pharmacokinetic Study of KX2 391 Ointment in Subj. w Actinic Keratosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Athenex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KX01-AK-01-US
Record Dates: First submitted 2015-01-05; First posted 2015-01-13 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2016-12

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- KX2-391 Ointment (Experimental)
  Interventions: Drug: KX2-391 Ointment

INTERVENTIONS:
Drug: KX2-391 Ointment — KX2-391 Ointment will be applied at a predetermined concentration to the treatment area for a predetermined time period.

SUMMARY:
This is a phase 1 study to access the safety and tolerability of KX2-391 ointment in subjects who have Actinic Keratosis. This study will also access the amount of KX2-391 drug that enters the blood stream through dermal application of the ointment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years old
2. Subject has a clinical diagnosis of stable, clinically typical AK
3. Subject has a treatment area on 1 dorsal forearm that in:

   Cohort 1:
   * Is one contiguous area
   * Measures 25 cm2
   * Contains 4 to 8 AK lesions that are clinically typical.

   Cohort 2:
   * Is one contiguous area
   * Measures 100 cm2
   * Contains 8 to 16 AK lesions that are clinically typical.
4. All women of childbearing potential (WOCBP) must be:

   * Post-menopausal, defined as at least 50 years of age with amenorrhea for at least 18 months, or
   * Surgically sterile, defined as having undergone a hysterectomy, bilateral oophorectomy or tubal ligation, or otherwise incapable of pregnancy.
   * Pre or perimenopausal and practicing a highly effective method of birth control, including hormonal prescription, oral contraceptives, contraceptive injections, contraceptive patch, and intrauterine device, for the duration of their participation in the study. Abstinence and double-barrier methods do not qualify as highly effective methods of birth control.
   * All woman of child-bearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test on Day 1 (Visit 2) prior to administration of KX2-391 Ointment dose.

   Contraception
   * Contraception must be consistently used for at least 3 months prior to screening to 3 months after the last KX2-391 Ointment dose.
   * Male Contraception: All men who are sexually active with female partners of child bearing potential must agree to ensure their partners use highly effective contraception and therefore will not father a child from screening to 3 months after the last dose of study medication.
   * Male and Female Contraception: All men and women subjects must agree to not donate sperm or eggs or attempt conception from screening to 3 months after the last KX2-391 Ointment dose.
5. Subject is, in the opinion of the investigator, in good general health based on medical history, physical examination, electrocardiogram (ECG), and clinical laboratory evaluations at screening.
6. Subject has clinically acceptable liver function at screening as demonstrated by:

   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2x upper limit of normal (ULN)
   * Total bilirubin ≤ ULN
7. No other screening laboratory test, including CBC results, considered clinically significant by the investigator
8. Subject is not lactating
9. Subject is willing and able to follow all study instructions and to attend all study visits
10. Subject is able to comprehend and willing to sign an Informed Consent Form (ICF)

Exclusion Criteria:

1. Subject has clinically atypical and/or rapidly changing AK lesions on the treatment area
2. Subject has current systemic malignancy
3. Subject has used any of the following systemic therapies within the specific period before Visit 1:

   * Retinoids; 180 days
   * Glucocortico-steroids; 28 days
   * Methotrexate or other anti-metabolites; 28 days
4. Subject has used any of the following topical therapies on the treatment area within the specified period before Visit 1:

   * Retinoids; 90 days
   * Glucocortico-steroids; 14 days
5. Subject has had any of the following of the AK therapies on the treatment area:

   Medical Therapies within 90 days (or until the site has healed, whichever is longer) before Visit 1:
   * Ingenol mebutate (eg, Picato)
   * 5-fluorouracil (eg, 5-FU; Efudex)
   * Imiquimod (eg, Aldara; Zyclara)
   * Diclofenac with or without hyaluronic acid (eg, Solaraze)
   * Moisturizer, emollients (12 hours prior to Visit 1)

   Surgical Modalities on the treatment area within 30 days (or until the site has healed following treatment, whichever is longer) before Visit 1:
   * Cryotherapy
   * Electrodesiccation
   * Laser, light (eg, photodynamic therapy, intense pulsed light) or any other energy based therapy
   * Chemical peels (eg, tricholoracetic acid)
   * Dermabrasion
   * Surgical removal (eg, curettage, excision)
6. Subject currently has, or has experienced any of the following on the treatment area within the specified period before Visit 1:

   * A cutaneous malignancy; 180 days
   * Sunburn; 28 days
   * Body art (eg, tattoo, piercing); currently
   * Excessive tan; currently
7. Subject has a history of sensitivity to any of the ingredients in the study medications
8. Subject is chronically taking a known strong inhibitor of CYP3A4
9. Subject has a skin disease (eg, atopic dermatitis, psoriasis, eczema) or condition (eg, scarring, open wounds) that, in the opinion of the investigator, might interfere with the study conduct or evaluations, or which exposes the subject to an unacceptable risk by study participation.
10. Subject has other significant uncontrolled or unstable medical diseases or conditions that, in the opinion of the investigator, would expose the patient to unacceptable risk from study participation.
11. Subject has participated in an investigational drug trial during which an investigational study medication was administered within 30 days before Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Overall safety and tolerability assessment as determined by laboratory, adverse event (AE) and serious adverse event (SAE) information. | 45 days
  Safety assessments will consist of determining and recording all AEs (including for both increasing and decreasing severity) and SAEs; laboratory evaluation for hematology, blood chemistry, and urine analytes; periodic measurement of vital signs and ECGs; and the performance of physical examinations as detailed in Table 3 of the protocol.
The amount of KX2-391 in the blood stream as determined by pharmacokinetic (PK) analysis: Cmax, Cmin, AUC0-t, AUC0-inf | 7 days
  Individual PK data will be listed by time. Cmax, Cmin, AUC0-t, AUC0-inf will be calculated for KX2-391 to determine systemic exposure.

SECONDARY OUTCOMES:
Actinic Keratosis (AK) lesion count | 45 days
  The AK lesion count is the investigator's assessment of the number of AK lesions in the treatment area.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Kramer, MD, Study Director — Kinex Pharmaceuticals
Locations (1):
- DermResearch, Inc., Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kempers S, DuBois J, Forman S, Poon A, Cutler E, Wang H, Cutler D, Fang J, Kwan R. Tirbanibulin Ointment 1% as a Novel Treatment for Actinic Keratosis: Phase 1 and 2 Results. J Drugs Dermatol. 2020 Nov 1;19(11):1093-1100. doi: 10.36849/JDD.2020.5576. PMID 33196758